CLINICAL TRIAL: NCT00801580
Title: Open Label, Non-randomized, Phase II Study on Fractioned Cyclophosphamide, Vincristine, Liposomal Doxorubicin or Doxorubicin, and Dexamethasone (MY HYPER-CVAD) in the Treatment of Relapsed Refractory Adult Acute Lymphoid Leukemia
Brief Title: My-HyperCVAD in the Treatment of Relapsed Refractory Adult Acute Lymphoid Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bologna (Other)
Responsible Party: Giovanni Martinelli, Institute of Hematology "L. & A. Seragnoli" - University of Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALL0206; Eudract: 2007-003884-30
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Lymphoid Leukemia
Keywords: relapsed ALL; refractory ALL; relapsed adult acute lymphoid leukemia
MeSH Terms: conditions — Leukemia, Lymphoid; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Doxorubicin

ARMS (1):
- 1 (Experimental): The patient receive 2 different drug combinations on this study. The first combination will consist of an intensive chemotherapy regimen (cyclophosphamide, mesna, methotrexate, doxorubicin liposomal or doxorubicin, vincristine, ARA-C (cytarabine) and dexamethasone). The second combination will consist of another intensive chemotherapy regimen (methotrexate and Ara-C [cytarabine]).
  Interventions: Drug: doxorubicin liposomal

INTERVENTIONS:
Drug: doxorubicin liposomal — * Cyclophosphamide
  * Mesna
  * Methotrexate
  * Doxorubicin liposomal
  * Vincristine
  * Dexamethasone
  * Rituximab
  * Cytarabine

SUMMARY:
The patient receive 2 different drug combinations on this study. The first combination will consist of an intensive chemotherapy regimen (cyclophosphamide, mesna, methotrexate, doxorubicin liposomal or doxorubicin, vincristine, ARA-C (cytarabine) and dexamethasone). The second combination will consist of another intensive chemotherapy regimen (methotrexate and Ara-C [cytarabine]).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALL (any type included), in patients who:

  * have relapsed after conventional chemotherapy* or,
  * are refractory to at least 1 cycle of chemotherapy*
* ECOG Performance score of 0-3
* Adequate hepatic and renal function, as defined by serum transaminases <2.5x ULN, bilirubin <1.5xULN, and creatinine <1.5x ULN.
* Age 18 years or greater.
* Documentation of written informed consent to participate in the trial.
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
* at least 3 weeks from prior chemotherapy or other investigational anticancer therapy with full recovery from prior toxicities.
* either men or women, accepting to practice effective contraception during the entire study period unless documentation of infertility exists.

Exclusion Criteria:

* Treatment with any investigational agent within 3 weeks prior to study therapy.
* Major surgeries within 4 weeks from study start or not fully recovered from any previous surgical procedure.
* Presence of any medical or psychiatric condition which may limit full compliance with the study or increase the risk associated with study participation or study drug administration, including but not limited to:

  * Presence of central nervous system (CNS) leukemia.
  * Active uncontrolled bacterial infection.
  * Known human immunodeficiency virus (HIV) infection.
  * Significant cardiovascular disease (i.e., uncontrolled arrhythmias, unstable angina), or a major thromboembolic event (myocardial infarction, stroke, transient ischemic attack, pulmonary embolism, or non-catheter-related deep-vein thrombosis) in the last 6 months.
  * Pregnancy or breast-feeding.
  * Malabsorption syndromes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Type, frequency, severity, timing and relatedness of adverse events (AE) | weekly
CR rate after any treatment cycle and at the end of the study | monthly

SECONDARY OUTCOMES:
The percentage of hematological responders after any treatment cycle | monthly
The percentage of cytogenetic and molecular responders after any treatment cycle in patients for whom genetic markers of minimal residual disease are available | monthly
Relapse free survival at month 6 and 12 | every 6 months
Overall survival at month 6 and 12 | every 6 months
The percentage of patients submitted to SCT after CR re-induction | every 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology "L. & A. Seragnoli", Bologna, Italy